CLINICAL TRIAL: NCT01663116
Title: "Phase Ib/IIa, Escalating Dose, Single Blind, Clinical Trial to Assess the Safety of the i.v Administration of Allogeneic Adipose-derived Mesenchymal Cells (eASCs) to Refractory Rheumatoid Arthritis (RA) Patients".
Brief Title: Cx611-0101, eASCs Intravenous Administration to Refractory Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cx611-0101
Record Dates: First submitted 2011-08-05; First posted 2012-08-13 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis Aggravated
Keywords: Rheumatoid arthritis; Expanded adipose derived allogeneic adult stem cells (eASCs)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): 1. first cohort: 1 million stem cells/kg administered at days 1, 8 and 15
  2. second cohort: 2 million stem cells / kg administered at days 1, 8 and 15
  3. third cohort: 4 million stem cells / kg administered at days 1, 8 and 15
  Interventions: Genetic: Stem cells
- Placebo (Placebo Comparator): Lactate Ringer´s solution
  Interventions: Genetic: Placebo

INTERVENTIONS:
Genetic: Stem cells — 1. first cohort: 1 million stem cells/kg administered at days 1, 8 and 15
  2. second cohort: 2 million stem cells / kg administered at days 1, 8 and 15
  3. third cohort: 4 million stem cells / kg administered at days 1, 8 and 15
  Arms: Treatment
Genetic: Placebo — 1. first cohort: 20 ml administered at days 1, 8 and 15
  2. second cohort: 40 ml administered at days 1, 8 and 15
  3. third cohort: 80 ml administered at days 1, 8 and 15
  Arms: Placebo

SUMMARY:
Phase Ib/IIa clinical trial of a new medicinal product of the somatic cell therapy class (eASCs). This study is designed as a multicenter, single blind, fixed dose escalation, with three treatment groups, controlled with placebo (randomization 3:1) whose target population are patients with rheumatoid arthritis refractory to at least two biologic.

DETAILED DESCRIPTION:
Traditionally, RA has been treated with non-steroidal anti-inflammatory drugs, glucocorticoids and non-biologics-DMARDs. Only non-biologics-DMARDs and, at a lesser extent, glucocorticoids have shown to be able to prevent or interrupt the inflammatory and destructive disease processes.

Mesenchymal stem cells (MSCs) are nonhematopoietic stromal cells that are able to differentiate into mesenchymal tissues such as bone, cartilage, muscle, ligament, tendon, and adipose. MSCs can be easily isolated from bone marrow or adipose tissue and rapidly expanded in culture. MSCs have also been shown to have immuno-suppressive and healing capacities, improve angiogenesis and prevent fibrosis. These properties could be used for novel therapeutic applications in various disorders, including rheumatoid arthritis, osteoarthritis (OA), genetic bone and cartilage disorders and bone metastasis. MSCs can potently modulate immune responses, showing antiproliferative and anti-inflammatory capacities.

This study is a multicenter phase Ib/IIa, escalating dose, single blind clinical trial to assess the safety of the intravenous administration of expanded allogeneic adipose-derived mesenchymal stem cells (eASCs) to refractory rheumatoid arthritis (RA) patients.

The primary objective of the study is to determine the safety, feasibility and tolerance, and to identify, if possible, the dose limiting toxicity (DLT) and the dose for future clinical trials on efficacy of the intravenous infusion of allogeneic eASCs for patients suffering rheumatoid arthritis (RA) under treatment with at least one non-biologic-Disease modifying antirheumatoid drug (DMARD) who have previously failed to treatment with at least two biologics. The secondary objective is to obtain information on the clinical and functional effects of the intravenous infusion of allogeneic eASCs in patients with RA and to explore pharmacodynamics parameters.

53 patients (i.e. patients having received at least one dose of study treatment) in three different cohorts are planned to be included in this clinical trial. Expansion will start after acute toxicity assessment of the first three patients of each cohort.

Dose and intervals for the trial consist of the following active groups: a) first cohort: 1 million cells/kg administered at days 1, 8 and 15; b) second cohort: 2 million cells / kg administered at days 1, 8 and 15; c) third cohort: 4 million cells / kg administered at days 1, 8 and 15.

ELIGIBILITY:
Inclusion criteria

Patients must meet all the following inclusion criteria to be eligible for study entry:

1. Must understand and voluntarily sign an informed consent form prior to the conduct of any study related assessment/procedures.
2. Subjects with RA under treatment with at least one non-biologic-DMARD and failure to treatment with at least two biologics.
3. Of either gender, aged ≥ 18 years at time of consent.
4. Able to adhere to the study visit schedule and other protocol requirements.
5. Have a diagnosis of RA for ≥6 months.
6. EULAR DAS28-ESR activity criteria >3.2.
7. Four tender joints to palpation and four swollen joints, based on a 68/66-joint count.
8. Be receiving treatment on an outpatient basis.
9. If taking methotrexate, leflunomide, or sulfasalazine, must have been treated for at least 16 weeks and on a stable dose (oral methotrexate ≤ 25 mg/week; parenteral methotrexate ≤ 20 mg/week; leflunomide ≤ 20 mg/day; sulfasalazine ≤ 3 g/day) for at least 4 weeks prior to the start of treatment and throughout the study. (See also section 7.5). The rest of the DMARDs (gold salts, etc) should be maintained at stable doses during at least the 4 weeks prior to the start of treatment and throughout the study (see also section 7.5).
10. If taking oral corticosteroids, must be on a stable dose of prednisone ≤ 10 mg/day or equivalent for at least 1 month prior to screening. ( See also section 7.5).
11. If taking NSAIDs, must be on stable dose for at least 2 weeks prior to screening and until they have completed the Week 24 study visit. (See also section 7.5).
12. Male subjects (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in activity in which conception is possible while on study medication and for at least 28 days after taking the last dose of study medication.
13. Females of Childbearing Potential* must have a negative urine pregnancy test at Screening and Baseline and must be willing to use one medically approved form of birth control when engaging in activity in which conception is possible while on study medication and for at least 28 days after taking the last dose of study medication.

    * A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral ovariectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).

Exclusion criteria

A patient CANNOT be recruited into this study if any of the following criteria is met:

1. Treatment with biologics within the following period prior to the start of treatment:

   1. Infliximab: 8 weeks
   2. Etanercept: 2 weeks
   3. Adalimumab and certolizumab: 4 weeks
   4. Abatacept, tocilizumab and golimumab: 8 weeks
   5. Rituximab: 6 months
   6. Anakinra: 3 days No treatment with biologics is allowed during the first 12 weeks after the start of the study treatment. Thus, the patients should have complied with the periods indicated above, and should not receive any biologics during the period specified.
2. Presence of a severe bleeding or thrombotic disorder.
3. History of known pulmonary embolism or known secondary anti-phospholipid syndrome.
4. Received any of the following treatments within 2 years prior to study entry: anti-cancer therapy (e.g. alkylating agents, anti-metabolites, purine analogues, monoclonal antibodies for malignancy).
5. Received within 4 weeks prior to the start of treatment: intra-articular, intramuscular or intravenous corticosteroids. (See also section 7.5).
6. Past or current malignant melanoma.
7. Past or current malignancy; except for in situ cervical cancer, non-invasive basal cell and squamous cell skin carcinoma, superficial bladder tumors (Ta and Tis) with a complete response duration of >10 years. In the case of lymphoma or breast cancer patients will be allowed to participate in the trial with a complete response duration of >20 years.
8. Other autoimmune diseases, previous or current inflammatory joint disease other than rheumatoid arthritis, currently active or previous recurrent bacterial, viral, fungal, or other infections including, but not limited to, tuberculosis and atypical mycobacterial disease, clinically significant abnormalities on chest radiograph, hepatitis B and C, and recurrent herpes zoster.
9. Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, Mycobacterium tuberculosis infection (TB) and active hepatitis B and C.

   For the screening of latent TB, the results of the tests performed in the last year according to the usual practice of the center or local guidelines will be accepted, as long as the investigator rules out a situation of high contact risk in the months after the last screening in accordance with the medical history of the patient.

   If the patient has a recent chest X-ray (performed in the month prior to enrollment in the study) and there is no clinical evidence or history suggestive of recent contact, it will not be necessary to repeat the test.
10. Subjects with signs of latent TB can be included if they have started treatment according to local guidelines at least one month prior to starting investigational therapy.
11. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months from screening, congestive heart failure of worse than grade II of the New York criteria.
12. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease.
13. History of significant cerebrovascular disease.
14. Subjects with congenital or acquired immunodeficiencies.
15. Known human immunodeficiency virus (HIV) positive.
16. Screening laboratory values (according to central laboratory):

    * Haemoglobin <5.6 mmol/L (9.0 g/dL).
    * Neutrophils <1.5 x 10(9)/L.
    * Leukocytes <3.0 x 10(9)/L.
    * Platelets <100 x 10(9)/L.
    * Serum IgG <lower limit of normal (LLN).
    * Alanine amino transferase (ALT) > 1.5 times the upper limit of normal (ULN).
    * Total bilirubin >2 mg/dl.
    * Aspartate amino transferase (AST) >1.5 times ULN.
    * Alkaline phosphatase (ALP) >2 times ULN.
    * Creatinine >133 mmol/L (1.5 mg/dL).
17. Serologic evidence of hepatitis C (HC) infection.
18. Serologic evidence of hepatitis B (HB) infection based on the results of testing for HBsAg, anti-HBc and anti-HBs antibodies as follows:

    * Subjects positive for HBsAg are excluded.
    * Subjects negative for HBsAg but positive for both anti-HBc and anti-HBs antibodies were eligible to participate.
    * Subjects negative for HBsAg and anti-HBc antibody but positive for anti-HBs antibody are eligible to participate.
    * Subjects negative for HBsAg and anti-HBs antibody but positive for anti-HBc antibody required clarification of their status by testing for HB DNA which if positive excludes the subject from participation.

      * Patients with documented vaccination against hepatitis B (primary and secondary immunization and booster) are considered negative.
19. Receipt of any vaccination (live, attenuated or killed) in 8 wks prior to baseline.
20. Subjects who had received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to screening.
21. Current participation in any other interventional clinical study.
22. Subjects known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
23. MRI is unfeasible, (e.g. due to the presence of pacemakers, hip replacements or severe claustrophobia).
24. Subjects with impossibility of having a radiological exploration.
25. Known allergies or hypersensitivity to antibiotics, HSA, DMEM, materials of bovine origin, gadolinium (MRI contrast) and Ringer's Lactate Solution.
26. Pregnancy and breastfeeding.
27. Any other condition which the PI judges would make patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events and Severe Adverse Events | 6 months follow up after the first administration
  Total number of Adverse Events and Severe Adverse Events, related and non-related with the medication will be recorded as a measure of tolerability and safety.

SECONDARY OUTCOMES:
Proportion of ACR20 patients/ACR50 patients/ACR70 patients (swollen joints*, tender joints**, physician global assessment***, patient global assessment***, patient´s assessment of pain ***, ESR/CRP, HAQ score) | At selection and screening visit, and once per month during 6 months after the last administration

CONTACTS AND LOCATIONS:
Overall Officials: José María Alvaro-Gracia, MD, PhD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (23):
- Spain (23):
  - Hospital General de Mérida, Mérida, Badajoz
  - Hospital U. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital U. de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario U. A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Clínico San Cecilio, Granada
  - Hospital U. Virgen de las Nieves, Granada
  - Hospital U. de Guadalajara, Guadalajara
  - Hospital de La Princesa, Madrid
  - Hospital U. Gregorio Marañon, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital U. La Paz, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital U. Marques de Valdecilla, Santander
  - Hospital Ntra. Sª de Valme, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital La Fe, Valencia
  - Hospital Dr. Peset, Valencia

REFERENCES:
- [Derived] Alvaro-Gracia JM, Jover JA, Garcia-Vicuna R, Carreno L, Alonso A, Marsal S, Blanco F, Martinez-Taboada VM, Taylor P, Martin-Martin C, DelaRosa O, Tagarro I, Diaz-Gonzalez F. Intravenous administration of expanded allogeneic adipose-derived mesenchymal stem cells in refractory rheumatoid arthritis (Cx611): results of a multicentre, dose escalation, randomised, single-blind, placebo-controlled phase Ib/IIa clinical trial. Ann Rheum Dis. 2017 Jan;76(1):196-202. doi: 10.1136/annrheumdis-2015-208918. Epub 2016 Jun 7. PMID 27269294